CLINICAL TRIAL: NCT00456209
Title: Lived Experiences of Adolescents in the Treatment Process of Cancer and the Impact of Occupations
Brief Title: Lived Experiences of Adolescents in the Treatment Process of Cancer and the Impact on Occupations
Status: Completed | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: 06.02.112
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Pediatric Cancer
Keywords: Lived Experiences; Adolescents; Cancer Treatment; Occupations
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this phenomenological study is to discover and illuminate the experiences of adolescents in the treatment process of cancer and the meanings they attach to these experiences, while maintaining their daily routines. The focus area of interest lies in the impact side-effects (psychological and physical) which these treatments may have on an individual's ability to participate with peers, maintain social activities, and be involved in daily occupation(s).

DETAILED DESCRIPTION:
This study will explore the following research questions: 1. How do adolescent patients in the treatment process of cancer perceive and describe their experience of engaging in occupational routines? 2. What effect does the treatment process of cancer have on an adolescent's ability to participate in life situations such as creating and maintaining relationships with family, friends, peers, students, or people with similar backgrounds?

By doing this study, researchers hope to gain information so that occupational therapists can increase the profession's present body of knowledge and better understand these individuals at a transitional period in their lives.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric cancer patients

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents being treating for cancer and the impact of their lived experience on engagement in occupations and social participation.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Lifestyle changes | 1 month
  Participants will be interviewed for observations of disease effect.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Grimaldi, MA, Principal Investigator
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States